CLINICAL TRIAL: NCT05629299
Title: Pilot Study to Detect Monkey Pox Virus in Sperm: POXSPERM
Acronym: POXSPERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0299; 2022-A01799-34 (Other: ID-RCB)
Record Dates: First submitted 2022-11-15; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Monkeypox
Keywords: Monkeypox Virus; semen; testicle; acute phase and follow-up
MeSH Terms: conditions — Mpox, Monkeypox | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monkey Pox infection (Other): Men will give semen, saliva, skin, urine and blood specimens
  Interventions: Biological: Samples

INTERVENTIONS:
Biological: Samples — Men will give semen, saliva, skin, urine and blood specimens

SUMMARY:
Given the current emerging epidemic of the MonkeyPox Virus (MPXV) and its route of transmission, the main objective of this pilot study is to characterize the presence of the MPXV in the semen of patients in the acute phase of infection and following this infection.

DETAILED DESCRIPTION:
Since May 2022, a total of 16 000 new cases of Monkey Pox Virus infection has been reported in 76 non-endemic countries. The WHO has declared this epidemic as a public health emergency. Principal routes of transmission are direct skin or mucosa contact or aerosol transmission. The current epidemic mainly affects men having sexual relations with others men and men reporting having recent sexual relations with new or multiple partners. We may wonder if there is a risk of transmission during an intercourse. Moreover, Monkey pox virus infection in human testicle has not been studied yet. Among viruses that infect human semen, some viruses can persist for several months or even years in the semen of cured men. In this context, we propose a research project about the pathophysiology of MPXV in the male genital tract by a clinical approach. Men with a diagnosis of MPXV infection confirmed by a positive PCR and who agreed to be included as volunteer will go to CECOS at Paule de Viguier Hospital, Purpan. Each patient will take a semen and urine sample, have a blood sample and a saliva sample, and a skin sample in case of a lesion; the earliest after the confirmation of the diagnosis of the infection (before the 7th day, the days will be noted) then on Day 15, Day 30, Day 60, Day 90 and Day 180.

ELIGIBILITY:
Inclusion Criteria:

* in the acute phase of MPXV infection and whose PCR reveals the viral genome in a skin sample or in any other sample.
* able to travel to the laboratory for the samples
* who gave his free and informed consent and having signed the consent
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Patient who has previously consulted for male infertility or who has previously performed an abnormal semen test (WHO standard)
* Patient with ejaculation disorder or unable to collect semen or with abnormal semen volume (<1.5 mL).
* Patient who presents serious clinical signs that do not allow him to travel to the investigation center.
* Patient under a protection regime (including guardianship, curatorship or safeguard of justice)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
MPXV genomic DNA | Day 0
  presence of MPXV DNA in the semen and others body fluids of infected patients in the acute phase and during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Manon CARLES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No